CLINICAL TRIAL: NCT06143917
Title: Efficacy of Parent-child Sleep Intervention to Improve Sleep Quality, Psychological Health, and Infant Health in Parents of Neonates.
Brief Title: Efficacy of Parent-child Sleep Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, VGHuser_Chien-Hui Chan, Principal investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-10-012C
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Sleep Quality; Psychological Health; Infant Health
Keywords: Parents; Neonate; Sleep education; Sleep quality; Psychological health; Infant health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parent-child sleep intervention (Experimental): Participants in the intervention will receive both the standardized usual care and parent-child sleep education, heart rate variability biofeedback training, and counseling and support.
  Interventions: Behavioral: parent-child sleep intervention
- Control (No Intervention): Participants in the control group will receive attention from the research nurse and the standardized usual care.

INTERVENTIONS:
Behavioral: parent-child sleep intervention — The intervention plan is as follows: (1) Parent-child sleep education includes two in-person session and four pre-recorded online sessions. Additionally, it provides educational handbooks tailored to the course content, segmented into sections for both parents and newborns. Each session lasts approximately 20 minutes; (2) Heart rate variability measurement and Heart rate variability biofeedback are conducted in classes in person. It guides parents through breathing exercises to activate the parasympathetic nervous system, thereby easing emotions and improving psychological health; (3) Professional counseling and support are provided separately at two weeks, one month, three months, and six months postpartum.
  Arms: parent-child sleep intervention

SUMMARY:
Background: Parents of healthy neonates commonly face sleep disruptions and disturbances after delivery. Notably, increasing challenges are evident among parents of ill infants who required clinical care after birth . These challenges can adversely affect psychological adaptation and parental efficacy which consequently impacting the infant's development. It is crucial to develop an effective parent-child sleep intervention for improving parent-infant sleep and mental well-being and uneventful family health outcomes.

Aim: To develop and evaluate the effects of parent-child sleep intervention on improving sleep quality, psychological health, and infant health in parents of infants at intermediate care nursery.

Methods: A randomized controlled trial will be conducted at the intermediate care nursery of a level III medical center at Taipei city. A total of 102 pairs of parents and infants will be recruited and randomly assigned to the experimental group or the control group. The intervention program consists of (1) parent-child sleep education, (2) heart rate variability biofeedback training, and (3) counseling and support. Data collection will be multiple time points, including baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum.

Anticipated results: Developing and evaluating a parent-child sleep intervention for postpartum parents and their infants. The findings will be an empirical evidence for pediatric care and family health promotion.

DETAILED DESCRIPTION:
The following measures will be used, including Insomnia Severity Index, Pittsburgh Sleep Quality Index, Brief Infant Sleep Questionnaire-Revised short form, Parental Efficacy Scale, State-Trait Anxiety Inventory, Infant Health Outcome Questionnaire. Objective data included actigraphy, and heart rate variability. Data will be analyzed using descriptive statistics and One-Way repeated measure ANOVA to examine the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18 years or older.
* Postpartum women with a singleton pregnancy, and the gestational age of their infant is at least 32 weeks.
* Postpartum women with a severe insomnia severity index score of ≥8 points.
* Postpartum women and their husbands or partners capable of reading, understanding, and communicating in Mandarin.
* Postpartum women and their husbands or partners with internet access and the ability to operate resources using a smartphone, tablet, or computer.
* Both postpartum women and their husbands or partners are willing to participate in the research process.

Exclusion Criteria:

* Postpartum women diagnosed with Insomnia Disorder, Anxiety Disorders, or Depression.
* Postpartum women suffering from arrhythmia or cardiovascular diseases.
* Postpartum women working in shifts.
* Infants with congenital abnormalities, neurological impairments (such as hydrocephalus, periventricular leukomalacia), requiring the use of tubes or respirators after discharge, or using medications that might affect sleep (such as caffeine, sedatives, muscle relaxant, anti-epileptic drugs, or pain medications).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-05-24 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in insomnia severity on the Chinese Version of the Insomnia Severity Index (ISI-C) at 1 month postpartum, 3 months postpartum, and 6 months postpartum | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  The ISI is a validated, self-reported questionnaire assessing insomnia severity over the past month period. Possible scores range from 0 (absence of insomnia) to 28 (severe insomnia).

SECONDARY OUTCOMES:
Change from Baseline in sleep quality on the Chinese Version of the Pittsburgh sleep quality index (PSQI-C) at 1 month postpartum, 3 months postpartum, and 6 months postpartum | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  PSQI-C is a validated, self-reported questionnaire assessing seven sleep quality components from 0 to 3, with a total score ranging from 0 (good sleep) to 21 (very poor sleep).
Change from Baseline in infant sleep quality on the Chinese Version of the Brief Infant Sleep Questionnaire-Revised Revised Short Form (BISQ-R-C SF) at 1 month postpartum, 3 months postpartum, and 6 months postpartum | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  BISQ-R-C SF is a validated questionnaire, the parents were instructed to refer to their child's sleep during the past week. Scores on each subscale and the total score are scaled from 0 to 100, with higher scores denoting better sleep quality, more positive perception of infant sleep, and parent behaviors that promote healthy and independent sleep.
Change from Baseline in anxiety symptoms on the Chinese Version of State-Trait Anxiety Inventory (STAI-C) at 1 month postpartum, 3 months postpartum, and 6 months postpartum | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  STAI-C is a validated, self-reported questionnaire assessing anxiety symptoms, total scores range from 20 to 80, with higher scores denoting a high level of anxiety.
Change from Baseline in parenting efficacy and satisfaction on the Chinese Version of the Parenting Sense of Competence Scale (PSOC-C) at 1 month postpartum, 3 months postpartum, and 6 months postpartum | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  PSOC-C is a validated, self-reported questionnaire assessing parenting self-efficacy, total scores range from 16 to 96, with higher scores denoting better perceived parental self-efficacy.
Infant health outcome | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  Infant health outcome will be measured using a structured questionnaire, including infant height, weight and feeding methods.
Satisfaction questionnaire | immediately after intervention
  Participants' satisfaction will be measured using a structured questionnaire.
Change from Baseline in heart rate variability (HRV) at 1 month postpartum, 3 months postpartum, and 6 months postpartum | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  Parents' heart rate variability will be measured using the professional version of the ''Eureka Destresser'' device produced by finesse technology co. ltd. This device has been approved by the National Communications Commission (NCC) and the Federal Communication Commission (Federal Communication). Commission, FCC) certification.
Activity and sleep monitor | Baseline, 1 month postpartum, 3 months postpartum, and 6 months postpartum
  Parents and infant sleep and daytime activity will be measured using ''ActiGraph GT9X Link'' to tracks sleep patterns, with recording 24-hour sleep diary.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hui Chan, Principal Investigator — Study Principal Investigator
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan